CLINICAL TRIAL: NCT00636402
Title: Vessel Sealing System Tonsillectomy vs Cold Knife Tonsillectomy: A Randomized, Paired Control Study of Efficacy and Adverse Effects
Brief Title: Study of Efficacy and Adverse Effects: Vessel Sealing System Tonsillectomy Versus Cold Knife Tonsillectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chulalongkorn University (Other)
Responsible Party: Assoc. Prof. Prakobkiat Hirunwiwatkul, Faculty of Medicine, Chulalongkorn University, Thailand
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENTCU_pkk2008_01
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2008-12-11 (Estimated); Status verified 2008-12

CONDITIONS: Tonsillitis; Obstructive Sleep Apnea
Keywords: Vessel Sealing System; Cold Knife; Tonsillectomy; Pain; Postoperative
MeSH Terms: conditions — Tonsillitis; Sleep Apnea, Obstructive; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Vessel Sealing System Tonsillectomy (VSST)
  Interventions: Procedure: Vessel Sealing System Tonsillectomy
- 2 (Active Comparator): Cold Knife Tonsillectomy (CKT)
  Interventions: Procedure: Cold Knife Tonsillectomy

INTERVENTIONS:
Procedure: Cold Knife Tonsillectomy — Cold Knife Tonsillectomy (CKT) will be done on the other side.
  Other Names: CKT
  Arms: 2
Procedure: Vessel Sealing System Tonsillectomy — Intervention by Vessel Sealing System Tonsillectomy (VSST) will be randomized and will be performed on one side.
  Other Names: VSST
  Arms: 1

SUMMARY:
This study was planned to compare vessel sealing system tonsillectomy (VSST) to the traditional cold knife tonsillectomy (CKT) with special regard to intraoperative bleeding, operative time, postoperative pain and hemorrhage.

DETAILED DESCRIPTION:
Tonsillectomy is one of the most common procedures performed by otolaryngologists. Intraoperative bleeding is a significant problem which requires hemostasis and causes prolonged operative time. Several different techniques are used to perform this operation. Efficacy in hemostasis and tissue trauma from different operative techniques may result in different operative time and different degrees of morbidity including intraoperative blood loss, postoperative pain and hemorrhage.

The vessel sealing system has been widely used in head and neck surgery because of its effectiveness and safety. It was also found quite effective and safe in tonsillectomy procedures, providing excellent hemostasis and minimal tissue trauma. This study was planned to compare vessel sealing system tonsillectomy (VSST) to the traditional cold knife tonsillectomy (CKT) with special regard to intraoperative bleeding, operative time, postoperative pain and hemorrhage.

Inclusion criteria are patients planned for tonsillectomy for indications of chronic tonsillitis or obstructive sleep apnea and written informed consent form is given from patient or patient's parents (in case of pediatric patient).

Exclusion criteria are pregnancy, history of bleeding disorders, unilateral tonsillectomy, much different size of both tonsils (If the difference is more than or equal to 2, it will be defined as much different in size in this study), patient unable to understand evaluation method or unable to be contacted via telephone. Outcome measurements are the following.

1. Operative time (minutes) will be started at the time of incision and ended at the time of complete hemostasis. After tonsillectomy on the first side is finished, 5-10 minutes is the lag time before tonsillectomy on the second side will be started in order to observe re-bleeding after operative time is recorded. If there is re-bleeding, the operative time will be changed and measured from the same starting time to the time of last complete hemostasis.
2. Amount of blood loss (milliliter) will be measured from amount of fluid including blood and saliva in the container and gauze. Measurement will be started at the time of incision and ended at the time of complete hemostasis in the same manner of operative time.
3. Pain score, postoperative hemorrhage or other adverse effects that the research assistant will record on post-op day 0-14 by using direct and telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* Patient planned for tonsillectomy for indications of chronic tonsillitis or obstructive sleep apnea
* Written informed consent form is given from patient or patient's parents (in case of pediatric patient)

Exclusion Criteria:

* Pregnancy
* History of bleeding disorders
* Unilateral tonsillectomy
* Much difference in size of both tonsils (if the difference is more than or equal to 2, it will be defined as much different in size in this study)
* Patient unable to understand evaluation method
* Patient unable to be contacted via telephone

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Intra-operative time | 1 day
Intra-operative blood loss | 1 day
Pain, postoperative | 14 days

SECONDARY OUTCOMES:
Postoperative bleeding and other adverse effects | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Prakobkiat Hirunwiwatkul, M.D., Principal Investigator — Faculty of Medicine, Chulalongkorn University, Thailand
Locations (1):
- Department of Otolaryngology, King Chulalongkorn Memorial Hospital, Bangkok, Bangkok, Thailand

REFERENCES:
- [Result] Lachanas VA, Hajiioannou JK, Karatzias GT, Filios D, Koutsias S, Mourgelas C. Comparison of LigaSure vessel sealing system, harmonic scalpel, and cold knife tonsillectomy. Otolaryngol Head Neck Surg. 2007 Sep;137(3):385-9. doi: 10.1016/j.otohns.2007.05.012. PMID 17765762
- [Result] Lachanas VA, Prokopakis EP, Bourolias CA, Karatzanis AD, Malandrakis SG, Helidonis ES, Velegrakis GA. Ligasure versus cold knife tonsillectomy. Laryngoscope. 2005 Sep;115(9):1591-4. doi: 10.1097/01.mlg.0000172044.57285.b6. PMID 16148700
- [Result] Prokopakis EP, Lachanas VA, Benakis AA, Helidonis ES, Velegrakis GA. Tonsillectomy using the Ligasure vessel sealing system. A preliminary report. Int J Pediatr Otorhinolaryngol. 2005 Sep;69(9):1183-6. doi: 10.1016/j.ijporl.2005.03.042. PMID 15961165
- [Result] Lister MT, Cunningham MJ, Benjamin B, Williams M, Tirrell A, Schaumberg DA, Hartnick CJ. Microdebrider tonsillotomy vs electrosurgical tonsillectomy: a randomized, double-blind, paired control study of postoperative pain. Arch Otolaryngol Head Neck Surg. 2006 Jun;132(6):599-604. doi: 10.1001/archotol.132.6.599. PMID 16785404
- [Result] Newman CJ, Lolekha R, Limkittikul K, Luangxay K, Chotpitayasunondh T, Chanthavanich P. A comparison of pain scales in Thai children. Arch Dis Child. 2005 Mar;90(3):269-70. doi: 10.1136/adc.2003.044404. PMID 15723913